CLINICAL TRIAL: NCT00157378
Title: Optimization of Acute Treatment in First Episode Schizophrenic Patients by New Pharmacological Treatments
Brief Title: Optimization of Acute Treatment in First Episode Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: Janssen-Cilag Ltd. (Industry); German Research Network On Schizophrenia (Network); Department of Psychiatry University of Bonn (Other); Heinrich-Heine University, Duesseldorf (Other); Department of Psychiatry University FU Berlin (Other); University of Göttingen (Other); University of Cologne (Other); Mainz University (Other); University Hospital Tuebingen (Other); Universität Duisburg-Essen (Other); University of Mannheim (Other); University of Jena (Other); Martin-Luther-Universität Halle-Wittenberg (Other); RWTH Aachen University (Other); University of Wuerzburg (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01GI9933-P2.1.2.1
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2000-01

CONDITIONS: Schizophrenia, First-Episode
Keywords: first episode,; schizophrenia,; atypical neuroleptics,; negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone; Haloperidol

INTERVENTIONS:
Drug: Risperidone, Haloperidol

SUMMARY:
The study is a multicenter, double-blind, randomized, parallel-group study with first episode schizophrenic patients. During a treatment phase of 8 weeks the patients are treated with Risperidone or Haloperidol. Aim of the project is to compare the effects of the atypical neuroleptic Risperidone with those of the conventional neuroleptic Haloperidol and to evaluate whether the assumed advantages of atypical neuroleptics compared to conventional neuroleptics are also present when both medications are administered in rather low daily dosages (min. 2 mg/d; max. 8 mg/d).

DETAILED DESCRIPTION:
Considering that first episode schizophrenic patients compared to multiple episode patients respond to lower dosages of neuroleptics, the study aims to reach neuroleptic response under the lowest possible dosage of the study medication (haloperidol or risperidone). Therefore the initial dosage of the study medication is 2 mg/d. Depending on the patients' symptomatology, the daily dosage of the study medication can be increased by 2 mg in weekly intervals up to a maximum dosage of 8 mg/d. Patients with the diagnosis of schizophrenia (F20, according to ICD-10-criteria) are consecutively enrolled in the study. The patients are assessed at weekly intervals during the acute inpatient treatment phase of 8 weeks. Apart from the weekly psychopathological characterisation additionally neuropsychobiological data are assessed at the time of admission and at the end of the study. Major questions of the study are, whether patients, who have been treated with risperidone compared with those, who have been treated with haloperidol show a better treatment outcome regarding negative symptoms and exhibit fewer extra-pyramidal motor side effects. Furthermore it is hypothesised, that the treatment with Risperidone has better effects on cognitive disorders/dysfunctions and depressive symptoms and that the patients, who receive Risperidone are more compliant and have a higher quality of life.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 criteria for first episode schizophrenia
* age between 18 and 55
* informed consent

Exclusion Criteria:

* legal reasons
* insufficient knowledge of the german language
* substance abuse or addiction
* pregnancy
* serious physical illness
* organic brain disease
* contraindication to neuroleptic treatment

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300
Dates: Start 2000-11; Study Completion 2004-12

PRIMARY OUTCOMES:
weekly assessment of psychopathology (e.g.PANSS)and side-effects

SECONDARY OUTCOMES:
cognitive disability
depression
life quality at time of admission & end of study

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Möller, Professor, Study Chair — Department of Psychiatry, Ludwig-Maximilians-University Munich
Locations (1):
- Department of Psychiatry, Ludwig-Maximilians-University, Munich, Germany

REFERENCES:
- See also: Related Info — http://www.kompetenznetz-schizophrenie.de/rdkns/325.htm